CLINICAL TRIAL: NCT01547182
Title: Cooperative Lifestyle Programs (CLIP-II)
Acronym: CLIP-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00018631; 2R18HL076441-06 (NIH)
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Cardiovascular Disease; Obesity; Physical Disability
MeSH Terms: conditions — Cardiovascular Diseases; Obesity | interventions — Caloric Restriction; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Weight Loss (Active Comparator): Caloric restriction
  Interventions: Behavioral: Caloric restriction
- Weight Loss and Aerobic Training (Experimental): Caloric restriction and walking
  Interventions: Behavioral: Caloric restriction; Behavioral: Aerobic Training
- Weight Loss and Resistance Training (Experimental): Caloric restriction and lifting weights
  Interventions: Behavioral: Caloric restriction; Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Caloric restriction — Caloric restriction
Behavioral: Aerobic Training — Walking
  Arms: Weight Loss and Aerobic Training
Behavioral: Resistance Training — Lifting weights
  Arms: Weight Loss and Resistance Training

SUMMARY:
The aim is to study the effects of weight loss and weight loss combined with different types of physical activity on changes in physical functioning of older adults who are at-risk for cardiovascular disease.

DETAILED DESCRIPTION:
Although aerobic exercise training (AT) has been the cornerstone of rehabilitation for patients with CVD or MetS, experts agree that with the escalating problem of obesity, prevention programs in this area need to target weight loss (WL) as well. This is reinforced by recent research of our own showing that obesity is a major risk factor for physical disability among older adults. From a translational perspective, clinical researchers have recommended that effective community partnerships are needed to deliver such programs. In response to this call, the investigators have recently completed a translational study funded by NHLBI, the Cooperative Lifestyle Intervention Program (CLIP). In this investigation, 288 obese, older adults with CVD or MetS were randomized to a successful aging control treatment (SA), AT, or AT+WL for 18-months. The primary outcome was mobility disability, assessed by performance on the 400 m Walk Test (400MWT), and our staff co-delivered the interventions with agents from 3 counties within the community infrastructure of North Carolina Cooperative Extension Centers. Whereas mobility improved significantly in the AT group compared to SA, AT+WL was superior to either SA or AT.

Building on CLIP, the investigators now propose to increase the translational significance of our interventions by having them delivered exclusively by community partners with our staff as "trainers and advisers" for desired behavior change. In addition, this study will provide the first large scale randomized controlled clinical trial to evaluate the effects of diet-induced weight loss (WL) on mobility in obese, older adults with CVD or the MetS as compared to WL combined with physical activity. The dual primary outcomes will be the 400MWT and muscle strength. Because uncertainty exists about the best approach for promoting WL in older adults due to concerns with the loss of lean mass, the design also permits a contrast between AT+WL and resistance exercise training (RT)+WL on muscle strength. Consistent with CLIP, our WL intervention will target a protein intake of 0.8 g∙kg body mass-1∙d-1. Reasons to consider RT+WL for older adults include: 1) the central role of muscle loss and decline in strength in mobility disability; 2) the underappreciated role of RT in cardiovascular health; 3) the influence of muscle mass on both resting and total energy expenditure as well as fat mass and bone health; and 5) the potential value of RT for improving mobility on tasks that depend heavily on the vertical movement of the center of mass (e.g., stair climbing). Eves and Plotnikoff22 have emphasized the importance of RT in older diseased populations and stated that "the investigators need to discover practical, sustainable, and economically viable ways to safely implement RT at the population level." To accomplish our goals, the investigators have created a community partnership with the YMCA, using 4 sites in Forsyth County, NC. One of the sites serves a large African American population. The investigators are moving this project from Cooperative Extension Centers to the YMCA because the former have neither the equipment nor the personnel necessary to independently train and monitor RT or AT.

ELIGIBILITY:
Inclusion Criteria:

* Residence: community-dwelling men and women from the counties of interest (SR)
* Age: between 60-79 yrs (SR)
* Activity Status: sedentary (less than 60 minutes of moderate intensity structured physical activity each week and occurs in no less than 10 minute blocks; SR)
* Adiposity: obese as defined by a BMI ≥ 30 (OAC)
* Medical Criteria: documented evidence of an MI, PCTI, chronic stable angina, cardiovascular surgery (coronary artery or valvular heart disease) or an ATP III diagnosis of the metabolic syndrome (PCP)
* Mobility Disability: disability defined as self-reported difficulty with walking ¼ mile, climbing stairs, lifting and carrying groceries, or performing other household chores such as cleaning and yard work (SR)
* Stability of Residence: does not plan to move out of the county of residence for the duration of the study (SR)
* Agreeableness: willing and able to participate in all aspects of the trial (SR)
* Consents: willing to give an informed consent and sign a HIPAA authorization form (SR)

Exclusion Criteria:

* Severe Symptomatic Heart Disease: evidence of unstable angina, symptomatic congestive heart failure, or exercise induced complex ventricular arrhythmias (PCP)
* MI or cardiovascular procedure within the last 3-months (PCP)
* Blood Pressure: a resting blood pressure > 160/100 mmHg (OAC)
* Severe Systemic Disease: diagnosis of Parkinson's disease, chronic liver disease (cirrhosis, chronic hepatitis, etc.), systemic rheumatic condition (rheumatoid arthritis, psoriatic arthritis, Reiter's disease, systemic lupus erythematosus, etc.), end stage renal disease or other systemic diseases or abnormal laboratory values which would preclude participants from safely participating in the protocol or impair their ability to complete the study (PCP)
* Cancer: active treatment for cancer other than non-melanotic skin cancer (PCP)
* Hearing or Sight Impairments: significant visual or hearing impairment that cannot be corrected and results in the inability to use the telephone or hear normal conversation (SR, OAC)
* Psychiatric Illness: bipolar depression or schizophrenia (defined as self-reported treatment for these conditions), currently receiving lithium or neuroleptics (PCP)
* Cognitive Impairment: dementia, delirium or impaired cognitive function as defined by a score on the Folstein Mini-Mental Status Exam < 21 (OAC)
* Participation in Other Trials: currently participating in or planning to participate in another medical intervention study (SR)
* Alcohol Intake: consuming more than 21 alcoholic drinks per week or alcoholism (SR)
* Functional Limitations: unable to walk unassisted (SR, OAC)
* English Literacy: unable to speak or read English
* Clinical Center Staff Evaluation: judged to be unsuitable for the trial for any reason by the clinic staff. A participant can be excluded prior to randomization because of some unspecified health problem that has been identified that would put the patient at risk for adherence or retention. These cases are discussed with a recruitment team consisting of the person who has raised the concern, an MD, and the study PIs.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2012-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
400-M walk test and Lower Leg Strength | 18 months

SECONDARY OUTCOMES:
CT Scan | November 2013-March 2017
  This study will generate preliminary estimates of the independent effects of exercise modality during weight loss on changes in CT-derived parameters of bone density and quality (i.e. structure, strength) and serum biomarkers of bone turnover in a subset (n=60) of CLIP II participants.

CONTACTS AND LOCATIONS:
Overall Officials: W. Jack Rejeski, PhD, Principal Investigator — Wake Forest University; Anthony Marsh, PhD, Principal Investigator — Wake Forest University
Locations (3):
- United States (3):
  - Kernersville YMCA., Kernersville, North Carolina
  - William G. White YMCA, Winston-Salem, North Carolina
  - Fulton YMCA, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rejeski JJ, Fanning J, Nicklas BJ, Rejeski WJ. Six-month changes in ghrelin and glucagon-like peptide-1 with weight loss are unrelated to long-term weight regain in obese older adults. Int J Obes (Lond). 2021 Apr;45(4):888-894. doi: 10.1038/s41366-021-00754-0. Epub 2021 Feb 1. PMID 33526855
- [Derived] Rejeski WJ, Marsh AP, Fanning J, Ambrosius WT, Walkup MP, Nicklas BJ. Dietary Weight Loss, Exercise, and Inflammation in Older Adults with Overweight or Obesity and Cardiometabolic Disease. Obesity (Silver Spring). 2019 Nov;27(11):1805-1811. doi: 10.1002/oby.22600. PMID 31689007
- [Derived] Kammire DE, Walkup MP, Ambrosius WT, Lenchik L, Shapses SA, Nicklas BJ, Houston DK, Marsh AP, Rejeski WJ, Beavers KM. Effect of Weight Change Following Intentional Weight Loss on Bone Health in Older Adults with Obesity. Obesity (Silver Spring). 2019 Nov;27(11):1839-1845. doi: 10.1002/oby.22604. Epub 2019 Sep 4. PMID 31486297
- [Derived] Beavers KM, Ambrosius WT, Rejeski WJ, Burdette JH, Walkup MP, Sheedy JL, Nesbit BA, Gaukstern JE, Nicklas BJ, Marsh AP. Effect of Exercise Type During Intentional Weight Loss on Body Composition in Older Adults with Obesity. Obesity (Silver Spring). 2017 Nov;25(11):1823-1829. doi: 10.1002/oby.21977. PMID 29086504
- [Derived] Marsh AP, Janssen JA, Ambrosius WT, Burdette JH, Gaukstern JE, Morgan AR, Nesbit BA, Paolini JB, Sheedy JL, Rejeski WJ. The Cooperative Lifestyle Intervention Program-II (CLIP-II): design and methods. Contemp Clin Trials. 2013 Nov;36(2):382-93. doi: 10.1016/j.cct.2013.08.006. Epub 2013 Aug 23. PMID 23974035